CLINICAL TRIAL: NCT06537843
Title: Safety and Efficacy of Venetoclax, Cytarabine and Metformin (VenCM) for Relapsed-Refractory and Induction-Ineligible Acute Myeloid Leukemia: Multicenter, Phase 2, Clinical Trial
Brief Title: Safety and Efficacy of Venetoclax, Cytarabine and Metformin (VenCM) for Relapsed-Refractory and Induction-Ineligible Acute Myeloid Leukemia
Acronym: VenCM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Municipal São José (Other)
Collaborators: Hospital de Clínicas da UFPR. Curitiba, PR, Brazil (Unknown); Hospital Ophir Loyola. Belem, PA, Brazil (Unknown); Hospital Universitario Polydoro Ernani de São Thiago. Florianopolis, SC, Brazil (Unknown); Hospital Amaral Carvalho. Jau, SP, Brazil (Unknown)
Responsible Party: Principal Investigator, Marcelo Pitombeira de Lacerda, MD, PhD, Hematology Specialist, Hospital Municipal São José
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VenCM-001
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Cytarabine; Metformin

STUDY DESIGN:
Intervention Model Description: Cohort 1: Newly diagnosed, induction-ineligible AML patients Cohort 2: Relapsed-refractory AML patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VenCM (Experimental): Venetoclax, Cytarabine, Metformin
  Interventions: Drug: Venetoclax; Drug: Cytarabine Injection; Drug: Metformin

INTERVENTIONS:
Drug: Venetoclax — Venetoclax, PO (tablet), 200 - 400mg, once-daily, 10 days per cycle (cycle 1), 5 days per cycle (cycle 2 and subsequent cycles).
Drug: Cytarabine Injection — Cytarabine, Subcutaneous injection, 10 - 100mg per square meter, once-daily, 10 days per cycle (cycle 1), 5 days per cycle (cycle 2 and subsequent cycles).
Drug: Metformin — Metformin, PO (tablet), 850mg, three times a day, 10 days per cycle (cycle 1), 5 days per cycle (cycle 2 and subsequent cycles).

SUMMARY:
Phase 2 clinical trial to evaluate the combination of venetoclax, cytarabine and metformin in relapsed-refractory and induction ineligible acute myeloid leukemia.

DETAILED DESCRIPTION:
Subjects will be included voluntarily after informed consent. Diagnosis of AML in accordance with the WHO classification and determination of inegibility to induction therapy or refractory or relapsed disease after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML in accordance with the World Health Organization criteria.
* Ineligibility for induction chemotherapy due to age (≥ 70 years) or, for patients 18 to 74 years of age, ECOG-PS 2 or 3, creatinine clearance below 60 mL/min/1,73m², left ventricular ejection fraction ≤ 50%.
* Projected life expectancy of at least 12 weeks.
* Not requiring supplemental oxygen or substitutive renal therapy.
* Female participants must be either postmenopausal, surgically sterile or practicing at least one protocol specified method of birth control starting at Study Day 1 through at least 180 days after the last dose of study drug.
* Male participants must agree, from Study Day 1 through at least 180 days after the last dose of study drug, to practice protocol specified methods of contraception and to refrain from sperm donation from initial study drug administration through at least 180 days after the last dose of study drug.
* Participant must voluntarily sign and date an informed consent form, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL).
* Known central nervous system (CNS) involvement with AML.
* Known human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection, or other active viral, bacterial or fungal infection requiring treatment.
* History of other malignancies prior to study entry, with the exception of non-melanoma skin cancer.
* Chronic Liver Disease and Cirrhosis with a class B or C Child-Pugh score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 12 months and 24 months
  Overall survival is defined as the time from patient inclusion to the date of death, using Kaplan-Meier methodology.

SECONDARY OUTCOMES:
Composite Complete Response Rate (CCR) | 12 months and 24 months
  Percentage of participants with complete remission (CR) or complete remission with partial (CRh) or incomplete blood count recovery (CRi) at any time during the study as assessed by the investigator. Response was based on physical examination, bone marrow results and hematology values according to the revised guidelines by the 2022 European LeukemiaNet AML Diagnosis and Treatment Recommendations.
Negative Measurable Residual Disease (MRD) Rate | 12 months and 24 months
  Percentage of participants with CR, CRh or CRi with negative measurable residual disease (MRD) as assessed by the investigator, in accordance with ELN recommendations, defined as having less than 10-³ residual blasts per leukocyte measured in the bone marrow.

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Hospital Ophir Loyola, Belém
  - Hospital de Clínicas da UFPR, Curitiba
  - Hospital Universitario Polydoro Ernani de Sao Thiago, Florianópolis
  - Hospital Amaral Carvalho, Jaú
  - Hospital Municipal Sao Jose, Joinville

IPD SHARING:
Plan to Share IPD: Undecided